CLINICAL TRIAL: NCT00002404
Title: The Effect of Treatment With Valacyclovir 500 mg BID on the Detection of HIV From Genital HSV Lesions in HIV-Infected Patients: A Double-Blind Crossover Study
Brief Title: The Effect of Valacyclovir on the Detection of HIV From Genital Herpes Lesions in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 291A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 1999-06

CONDITIONS: Herpes Simplex; HIV Infections
Keywords: HIV-1; Antiviral Agents; Herpes Genitalis; Recurrence; DNA, Viral; RNA, Viral; valacyclovir; Herpesvirus 2, Human
MeSH Terms: conditions — Herpes Simplex; HIV Infections; Herpes Genitalis; Recurrence | interventions — Valacyclovir

INTERVENTIONS:
Drug: Valacyclovir hydrochloride

SUMMARY:
The purpose of this study is to see if valacyclovir affects the detection of HIV in genital herpes lesions in HIV-infected patients. Valacyclovir is used to treat recurrent genital herpes.

DETAILED DESCRIPTION:
Following evaluation for 2 consecutive episodes of genital herpes in this double-blind, crossover study, 30 HIV-1 positive patients are randomized to receive either valacyclovir or placebo.

All patients are treated for 10 days.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Serologically documented HSV-2 and HIV-1 infection.
* History of recurrent genital herpes that presents at least 3 recurrences within the 12 months prior to the start of study.
* No contraindications to valacyclovir.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

1. Hepatic impairment.
2. Impaired renal function (creatinine above 2 mg/dl).
3. Malabsorption syndrome or other gastrointestinal dysfunction.
4. Any other condition that in the investigator's opinion would interfere with study procedures or successful completion of protocol.

Patients with the following prior conditions are excluded:

History of hypersensitivity to acyclovir or valacyclovir.

Prior Medication:

Excluded:

* Participation in any investigational drug trial within 1 month prior to entry on study.
* Systemic anti-HSV therapy within 7 days prior to start of study drug.

  1. Probenecid.
* Suppressive treatment with medication that has anti-HSV activity.

Required:

- Stable antiretroviral therapy or no therapy for at least 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30